CLINICAL TRIAL: NCT05774652
Title: LiPO Teen (the Lifestyle in Pregnancy and Offspring Teenagers): Identification of Modifiable Risk Factors for Childhood Obesity - a Follow-up of a Randomized Controlled Trial
Brief Title: LiPO Teen (the Lifestyle in Pregnancy and Offspring Teenagers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Steno Diabetes Center Odense (Other); University of Southern Denmark (Other); Statens Serum Institut (Other); University of Aarhus (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Birgitte Moeller Luef, M.D, Ph.D Student, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LiPO-Teen
Record Dates: First submitted 2023-02-16; First posted 2023-03-20 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Life Style, Healthy; Follow-up; Gestational Weight Gain; Body Weight
MeSH Terms: conditions — Obesity; Gestational Weight Gain; Body Weight

STUDY DESIGN:
Intervention Model Description: The objective of the LiPO-Teen project is to perform a clinical follow-up study of the eligible 301 mothers who completed the trial until delivery with a liveborn child, and their 14 year-old offspring.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet + physical activity (Experimental): Diet + physical activity Dietary advise and advise on physical activity
  Interventions: Behavioral: Lifestyle intervention Dietary advise and/or advise on physical activity
- Control group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Lifestyle intervention Dietary advise and/or advise on physical activity — Lifestyle intervention Dietary advise and/or advise on physical activity
  Arms: Diet + physical activity

SUMMARY:
The study is a follow-up of a Randomized Controlled Trial (RCT) performed in 2007-10 - the "Lifestyle in Pregnancy" LiP study.

The LiP study included 360 pregnant women with BMI ≥30 kg/m2 from Odense University Hospital and Aarhus University Hospital. The women were randomized to intervention with low-calorie diet and physical activity from gestational age 10-14 in pregnancy and until delivery - or to a standard care control group. The objective of the LiPO-Teen project is to perform a clinical follow-up study of the eligible 301 mothers who completed the trial until delivery with a liveborn child, and their 14 year-old offspring. The overall ambition is to understand whether lifestyle intervention in pregnancy prevents obesity and its complications across generations, with a specific focus on modifiable factors.

DETAILED DESCRIPTION:
LiPO Teen (the Lifestyle in Pregnancy and Offspring Teenagers): Identification of modifiable risk factors for childhood obesity - a follow-up of a randomized controlled trial.

The objective of the LiPO-Teen project is to perform a clinical follow-up study of the eligible 301 mothers who completed the trial until delivery with a liveborn child, and their 14 year-old offspring.

In the original trial women were randomized 1:1 to intervention or control. The participants (both mother and child in pair) who completed the initial LiP study will be invited to a 2-hour examination now 14 years after the intervention during pregnancy to evaluate the effect of the intervention on both mother and child long term.

ELIGIBILITY:
Inclusion Criteria:

* Mothers in the initial LiP study selected at the baseline study in 2007-2010
* Teenagers of mothers in the initial LiP study

Exclusion Criteria:

• None

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 301 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Fat mass index , measured by DEXA scan. | 2 years data collection
  Body composition Assessed by Dual-Energy X-ray Absorptiometry (DEXA). Hologic Horizon, serie number: 301872M. Fat mass, lean mass and bone density will be calculated.
  Fat mass index in both mothers and offspring (Fat mass index (FMI) defined as: FM (kg) / height (m)2).

SECONDARY OUTCOMES:
Glycemic variability | 2 years data collection
  Continuous glucose monitoring (CGM, DEXCOM G6Pro): 10 days recording of fasting glucose and postprandial glucose values. Glucose variability will be assessed using a device, which performs repeated glucose measurements in the skin providing insights into glucose fluctuations throughout the day and night.
Mental health | 2 years data collection
  Assessed by questionnaires, validated to mother and child respectively
Diet composition | 2 years data collection
  Assessed by FFQ (food frequency questionnaire), validated to mother and child respectively
Physical activity (PA) | 2 years data collection
  Pattern and level of PA will be measured 7 days (24/7) monitored by activity tracker on the wrist (Actigraph GT3X+).
Puberty stage | 2 years data collection
  According to the classifications of Marshall and Tanner
Blood pressure | 2 years data collection
  Standardized sitting measurement, average of 3 measures. Both systolic and diastolic blood pressure will be measured.
Epigenetic examinations | 2 years data collection
  Blood samples:
  The epigenetic profile of DNA samples extracted from whole blood will be characterized by Genome-wide DNA methylation using Infinium MethylationEPIC v2.0 Kit. Principle component and hierarchical clustering analyses will be used to identify associations between methylation patterns and a range of clinical characteristics, biomarkers as well as gene expression levels (RNAseq).
Metabolic and inflammatory markers | 2 years data collection
  Blood samples: Glucose
HbA1c | 2 years data collection
  Blood samples: HbA1c
Metabolic markers | 2 years data collection
  Blood samples: Lipids (total cholesterol, HDL, LDL, triglyceride)
Electrolytes | 2 years data collection
  Blood sample: Electrolytes
Insulin | 2 years data collection
  Blood sample: Insulin
Vitamin D | 2 years data collection
  Blood sample: Vitamin D
Selenium | 2 years data collection
  Blood sample: Selenium
Zinc. | 2 years data collection
  Blood sample: Zinc
C-peptide | 2 years data collection
  Blood sample: C-peptid
Leptin | 2 years data collection
  Blood sample: Leptin
Adiponectin | 2 years data collection
  Blood sample: Adiponectin.
HsCRP. | 2 years data collection
  Blood sample: HsCRP.
IL6 | 2 years data collection
  Blood sample: IL6
Ferritin | 2 years data collection
  Blood sample: Ferritin
Leukocytes | 2 years data collection
  Blood sample: Leukocytes
Kidney function (e-GFR) | 2 years data collection
  Blood sample: Kidney function (e-GFR)
Liver enzymes | 2 years data collection
  Blood sample: Liver enzymes

CONTACTS AND LOCATIONS:
Overall Officials: Christina A Vinter, M.D. Ph.D., Principal Investigator — Department of Gynecology and Obstetrics. Odense University Hospital. University of Southern Denmark
Locations (1):
- Steno Diabetes Center Odense, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luef BM, Jensen NH, Knorr S, Kristensen K, Overgaard M, Stentebjerg LL, Catalano PM, Moller S, Maindal HT, Jensen DM, Vinter CA. Study protocol for a 15-year follow-up of a randomized controlled trial on lifestyle intervention in pregnancy: assessing long-term effects on body composition, metabolic traits, and mental health in mothers and offspring. Trials. 2026 Jan 14. doi: 10.1186/s13063-025-09418-0. Online ahead of print. PMID 41535891